CLINICAL TRIAL: NCT05676905
Title: Prospective Multicenter Observational Study on the Use of NEOCEMENT® for the Treatment of Bone Defects
Status: Terminated | Type: Observational
Why Stopped: The study was terminated following a change in company management.
Sponsor: Bioceramed (Industry)
Collaborators: European Clinical Research Infrastructure Network (Other); Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: TBMED1.1
Record Dates: First submitted 2022-11-28; First posted 2023-01-09 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-11

CONDITIONS: Bone Deformity
Keywords: Bone cement; Observational study; Real-world study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Neocement — Bone graft substitutes
  Other Names: Neocement Inject P

SUMMARY:
Neocement is a CE marked device, registered in INFARMED (Portuguese National Competent Authority) and Department of Planning and Organisation of the National Health Service - General board of Medical Devices, pharmaceutical services, and safety in healthcare (Italy). This protocol does not include any new intended uses, new populations, new materials or design changes.

DETAILED DESCRIPTION:
Neocement developed by Bioceramed is a calcium phosphate cement, composed of a liquid and a solid phase that upon mixing form a mouldable paste which hardens within 4-8 minutes due to an isothermal reaction.

This device is intended to be used in filling bony voids or gaps in the extremities, which have either been surgically created, or the result of traumatic injury to the bone and are not intrinsic to the stability of the bony structure. Hence, it is intended to be used by healthcare professionals (surgeons) when bone ingrowth and consolidation are required.

Neocement is contraindicated to use in load bearing applications, and must not be used where the implantation site is unstable and not rigidly fixed. Additionally, it is also not indicated to use in cases where the implantation site presents infection, nor in cases where poor bone healing would be expected, such as metabolic, immunologic or systemic disorders.

Bone grafting technique has been employed for several decades by orthopaedic surgeons to potentiate the process of bone repair across all orthopaedics' subspecialties.

Despite autografts with cancellous bone being considered the "gold standard" for bone regeneration due to their osteogenic elements, there are numerous disadvantages associated to this technique, including extended surgical time, local pain and swelling from donor segments.

The use of synthetic substitutes, like calcium phosphate cements, have significant advantages, including decreased risk of infection from human pathogens, and unlimited availability in various shapes and sizes. Thus, reconstruction and/or filling of bone defects caused by trauma, disease, or tumour resection in long bones using calcium phosphate cements has proven to be an effective and safe alternative to reduce donor-site morbidity associated to autografting, whilst providing support for bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bone defect treatment who meet predefined criteria in Instructions For Use (IFU) of Neocement® / Neocement® Inject P.
* Age ≥ 18 years of both genders (male and female)
* Patient signed informed consent form (for data collection)
* Bone defects surgically created or osseous defects created from traumatic injury to the bone
* Bone skeletal defects that are not intrinsic to the stability of bone structure OR site which can be stabilized

Exclusion Criteria:

* Acute or chronic infection at the surgical site;
* Metabolic bone diseases;
* Severe degenerative disease conditions in which general bone grafting is not advisable;
* Active malignancy.
* Inability to understand consent and objectives of the study;
* Pregnant women or breastfeeding women;
* Unable to undergo medical monitoring for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone graft substitute patients who underwent surgery with Neocement and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Bone consolidation (Neer/ RUST classification) | 24 months
  Neer classification is used for trabecular bone:
  Healed: Cyst filled by new bone, with or without small radiolucent area(s) < 1 cm in size
  Healing with defects: Radiolucent area(s) < 50% of the diameter of bone, with enough cortical thickness to prevent fracture
  Persistent cyst: Radiolucent area > 50% of diameter of the bone and with a thin cortical rim. No increase in the size of the cyst.
  Recurrent cyst: Cyst reappeared in a previously obliterated area, or a residual radiolucent area has increased in size)
  RUST is classified according to the scores:
  Score 1: Fracture Line, No Callus
  Score 2: Fracture Line, Visible Callus
  Score 3: Fracture Line, Bridging Callus
  Score 4: No fracture line, remodelled

SECONDARY OUTCOMES:
Functional scores | 24 months
  Functional scores are classified as Hip disability and Osteoarthritis Outcome Score, Knee disability and Osteoarthritis Outcome Score, Foot and Ankle Ability Measure, where 0 points is the worst possible score and 100 points is the best possible score.

OTHER OUTCOMES:
Adverse events | 24 months
  Assess patients' health during recovery
Quality of life measured through the SF-36 Questionnaire | 24 months
  Collect usability feedback on the device
Technical success rate | 24 months
  Successful delivery of the bone substitute in the bone defect

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Ribeiro, M. Doctor, Study Chair — Hospital Lusíadas Lisboa
Locations (1):
- Centro Hospitalar Universitário de Lisboa Central, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No